CLINICAL TRIAL: NCT05679700
Title: The Effect of Rigid Taping in Chronic Stroke Patients With Knee Hyperextension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Suleyman Korkusuz, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA-22045
Record Dates: First submitted 2022-12-21; First posted 2023-01-11 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Chronic Stroke
Keywords: Gait Analysis; Stroke; Knee Hyperextension; Rigid Taping
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic stroke patients with knee hyperextension (Experimental)
  Interventions: Other: Rigid Taping

INTERVENTIONS:
Other: Rigid Taping — Rigid taping was applied to stroke patients with knee hyperextension.

SUMMARY:
In this study, it is aimed to examine the effect of rigid taping on hyperextension control in stroke patients with knee hyperextension in the stance phase of gait.

Hypothesis Ho: Rigid taping has no effect on the control of knee hyperextension in stroke patients.

H1: Rigid taping has an effect on the control of knee hyperextension in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke at least 6 months ago
* Ambulation with or without a walking aid (walker, cane or tripod)
* To be between 0-3 points according to the Modified Rankin Scoring
* Presence of spasticity in any of the lower extremity muscles with a value of at least 1 according to the Modified Ashworth Scale
* Getting a score of 24 or higher on the Mini Mental Test
* Presence of hyperextension in the stance phase of gait

Exclusion Criteria:

* Having more than one stroke history
* Being diagnosed with dementia
* Having a previous diagnosis of orthopedic, psychiatric or other neurological disease
* Having a situation that prevents communication
* History of surgery or joint contracture involving the lower extremities and gait

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2023-10-11 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Vicon Motion Capture System | Baseline
  A total of 16 reflective signs will be placed on certain anatomical points of the participants. Gait analysis will be performed at a distance of 5 meters from the participants. The three-dimensional positions of the reflective marks will be recorded with the 8-camera Vicon motion capture system.
Blade Software System | Baseline
  Data obtained from Vicon motion capture system will be processed with Blade software. With the blade software, kinematic data will be obtained in the computer environment.

CONTACTS AND LOCATIONS:
Overall Officials: Kadriye Armutlu, Prof. Dr., Study Chair — Hacettepe University; Süleyman Korkusuz, MSc, Principal Investigator — Hacettepe University; Mehmet Akif Topçuoğlu, Prof. Dr., Study Chair — Hacettepe University; Serdar Arıtan, Asst.Prof, Study Chair — Hacettepe University; Nihat Özgören, MSc, Study Chair — Hacettepe University; Ali Naim Ceren, Msc, Study Chair — Hacettepe University
Locations (1):
- Hacettepe University, Altındağ, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper A, Alghamdi GA, Alghamdi MA, Altowaijri A, Richardson S. The relationship of lower limb muscle strength and knee joint hyperextension during the stance phase of gait in hemiparetic stroke patients. Physiother Res Int. 2012 Sep;17(3):150-6. doi: 10.1002/pri.528. Epub 2011 Dec 7. PMID 22147298
- [Background] Geerars M, Minnaar-van der Feen N, Huisstede BMA. Treatment of knee hyperextension in post-stroke gait. A systematic review. Gait Posture. 2022 Jan;91:137-148. doi: 10.1016/j.gaitpost.2021.08.016. Epub 2021 Aug 24. PMID 34695721
- [Derived] Korkusuz S, Korkusuz BS, Ozgoren N, Aritan S, Ceren AN, Topcuoglu MA, Balkan AF. Knee hyperextension in chronic stroke: Associated biomechanical and neuromuscular factors. Clin Biomech (Bristol). 2025 Aug;128:106617. doi: 10.1016/j.clinbiomech.2025.106617. Epub 2025 Jul 17. PMID 40706550